CLINICAL TRIAL: NCT02903173
Title: An Observational Study of Post-cesarean Delivery Respiratory Patterns Using a Non-invasive Minute Ventilation Monitor (Exspiron ™ System)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Respiratory Motion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00057206
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy; Analgesia; Respiratory Depression; Obstructive Sleep Apnea; Postpartum
Keywords: respiratory depression; postpartum; neuraxial morphine; cesarean delivery
MeSH Terms: conditions — Agnosia; Respiratory Insufficiency; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women who undergo cesarean delivery

SUMMARY:
The purpose of this study is to evaluate the breathing patterns of women who undergo cesarean delivery with spinal or epidural morphine for post-operative pain control in the first day after surgery. Some women who undergo cesarean delivery may be at risk for respiratory complications related to opiate administration for post-operative pain. The primary aim of this study is to evaluate post-operative minute ventilation in women who undergo cesarean delivery using a novel method of non-invasive minute ventilation monitoring, and to see if there are predictive risk factors that may predispose women to post-operative hypoventilation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* planned cesarean delivery with neuraxial morphine for post-operative analgesia

Exclusion Criteria:

* Non-English speaking subjects
* patients who undergo urgent or emergent cesarean deliveries
* patients who receive general anesthesia or do not receive neuraxial morphine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be pregnant woman recruited from the Duke Birthing Center (DBC) in the 5700 unit of Duke Hospital who are scheduled for planned cesarean delivery.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-02; Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Change in minute ventilation | baseline and 24 hours post cesarian delivery

SECONDARY OUTCOMES:
Berlin Questionnaire | Baseline
STOP-BANG Questionnaire | Baseline
Epworth Sleepiness Scale | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dominguez, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided